CLINICAL TRIAL: NCT05101499
Title: Randomized Study on Akin Osteotomy: Fixation Versus Non-fixation
Brief Title: Study on Akin Osteotomy: Fixation Versus Non-fixation (Fixakin)
Acronym: Fixakin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Clinique Blomet (Unknown); European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A00717-48
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Akin Osteotomy; Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AKIN osteotomy with screw fixation (Experimental)
  Interventions: Procedure: AKIN osteotomy with screw fixation
- AKIN osteotomy without screw fixation (Active Comparator)
  Interventions: Procedure: AKIN osteotomy without screw fixation

INTERVENTIONS:
Procedure: AKIN osteotomy with screw fixation — A simple skin speck is made on the medial aspect of the hallux, in the metaphyseal area, using a 3 mm beaver blade. The tissue is lifted from the bone using an elevator medially and dorsally on the phalanx. A Shannon 2x12 mm burr is then positioned transversely by making the osteotomy which must preserve a lateral hinge, a guarantee of stability in the event of non-fixation.
  Fixation with a screw will be effected by another skin speckle allowing access to the infero-medial area of the phalangeal base. A pre-hole can be made with the same bur to facilitate the introduction of the guide wire for osteosynthesis, which is not specific.
  Arms: AKIN osteotomy with screw fixation
Procedure: AKIN osteotomy without screw fixation — This is the same procedure as the procedure under study, without the fixation by a target: a simple skin speck is performed on the medial face of the hallux, in the metaphyseal area using a beaver blade. of 3 mm. The tissue is lifted from the bone using an elevator medially and dorsally on the phalanx. A Shannon 2x12 mm burr is then positioned transversely by making the osteotomy which must preserve a lateral hinge, a guarantee of stability in the event of non-fixation.
  Arms: AKIN osteotomy without screw fixation

SUMMARY:
We hypothesize that the Akin screw fixation osteotomy technique provides better postoperative mobility of the metatarsophalangeal hallux joint compared to the non-fixation technique.

DETAILED DESCRIPTION:
Compare the screw fixation technique of Akin's osteotomy, compared to the technique without fixation, on the postoperative mobility of the metatarsophalangeal joint of the hallux at one year postoperatively in patients ( patients operated on for an isolated hallux valgus, that is to say without any associated lateral movement, by percutaneous technique (MICA or PERC).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years-old
* Patient undergoing percutaneous surgery for Hallux valgus with first hybrid and / or percutaneous ray procedure without rotation disorder,
* First line surgery,
* Absence of metatarsophalangeal osteoarthritis,
* Persistence of mobility of the hallux metatarsophalangeal gland,
* Subject benefiting from a social protection insurance
* Patient having signed the free and informed consent / Patient having given his express consent / Patient having been informed and not opposing this research.

Exclusion Criteria:

* Rotation disorder,
* Rheumatoid foot,
* Hallux rigidus.
* Patient participating in another clinical study
* Minors:
* Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision;
* Pregnant, breastfeeding or parturient woman;
* Hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2021-11-18 (Estimated)

PRIMARY OUTCOMES:
Overall mobility of the metatarsophalangeal hallux joint in degre | 1 year
  Overall mobility of the metatarsophalangeal hallux joint in degree, one year after surgery, measured by a goniometer, as the amplitude between plantar flexion and dorsiflexion.

CONTACTS AND LOCATIONS:
Locations (1):
- BLOMET clinic, Paris, IDF, France